CLINICAL TRIAL: NCT01875029
Title: The Effects of Transcranial Direct Current Stimulation (tDCS)Combined With Back School in Subjects With Chronic Low Back Pain. Randomised Control Trial Study.
Brief Title: tDCS Effects on Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, MD, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Low Back Pain_tDCS
Record Dates: First submitted 2013-05-21; First posted 2013-06-11 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Low Back Pain; Chronic Pain
Keywords: Low back pain; chronic pain; tDCS; transcranial direct current stimulation
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sham-tDCS + Back School (Sham Comparator): This group will receive sham-tDCS for 5 days before back school beginning. The anode will be placed on the primary motor cortex (M1) of the dominant hemisphere and the cathode on the contralateral supraorbital area. The direct current is transmitted through a pair of sponge electrodes, with a surface of 35 cm2 (7x5), soaked in saline solution and, it is generated by a constant current stimulator, with rechargeable batteries. This continuous stimulation lasted 30 seconds, with an intensity of 1 milliampere.
  The back school session, a behavioural intervention,will be given 10 times for 4 weeks.
  Interventions: Device: sham-tDCS + back school
- real-tDCS + Back School (Experimental): This group will receive continuous stimulation lasting 20 minutes daily, for 5 days before back school beginning. The back school session, a behavioural intervention,will be given 10 times for 4 weeks.
  Transcranial direct current stimulation (tDCS) will be administered as follows. The anode will be placed on the primary motor cortex (M1) of the dominant hemisphere and the cathode on the contralateral supraorbital area. The direct current is transmitted through a pair of sponge electrodes, with a surface of 35 cm2 (7x5), soaked in saline solution and, it is generated by a constant current stimulator, with rechargeable batteries. This continuous stimulation lasted 20 minutes, with an intensity of 1 milliampere.
  Interventions: Device: real-tDCS + back school

INTERVENTIONS:
Device: sham-tDCS + back school — sham tDCS + back school
  Arms: sham-tDCS + Back School
Device: real-tDCS + back school — real tDCS + back school
  Arms: real-tDCS + Back School

SUMMARY:
Back School (BS) is a behavioural intervention designed to treat and prevent chronic low back pain. Up to date clinical research studies have shown that transcranial direct current stimulation (tDCS) is able to decrease the intensity and duration of pain modulating the activity of brain areas involved in the circuits that regulate pain and facilitating the mechanisms inhibitors descendants of pain control.

The aim of this study is to test the feasibility of combining tDCS with a behavioural intervention (i.e. BS) in subjects with chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain involves high individual and social costs. Back School (BS) is a behavioural intervention designed to treat and prevent the aforementioned condition. Up to date clinical research studies have shown that transcranial direct current stimulation (tDCS) can be considered a reliable tool for chronic pain. It has been shown how tDCS is able to decrease the intensity and duration of pain modulating the activity of brain areas involved in the circuits that regulate pain, such as the thalamus, and facilitating the mechanisms inhibitors descendants of pain control. The aim of this study is to test the feasibility of combining tDCS with a behavioural intervention (i.e. BS) in subjects with chronic low back pain. Specifically, we will test their effects on low back pain intensity and participation of patients' in daily activities.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged > 18 years and <75 years
* presence of non-specific chronic low back pain diagnosed > 2 years
* presence of a chronic pain measurable with the VAS scale not less than 3 during a 2 weeks daily VAS monitoring
* pain refractory to drugs (opioid analgesics, tricyclic antidepressants, antiepileptic drugs). It is considered a refractory pain if there is at least 6 months of treatment with at least 2/3 of the above drugs

Exclusion Criteria:

* spine surgery
* cognitive impairment assessed with Mini Mental Status Examination <24
* contraindications to tDCS: presence of a history of epilepsy, frequent headaches or neck pain, implantable devices (ventriculoperitoneal shunts, pacemakers, intrathecal pumps, intracranial metal implants)
* Contraindications to tDCS: intracranial metal implants that can be stimulated, incorrectly positioned or over-heated by the electric current
* Neurological or psychiatric pathology
* severe cardio-pulmonary, renal, hepatic diseases
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Visual Analogue Scale (VAS) for pain | 1)one day pre-tDCS treatment. 2) Every day, for 5 days pre and post 20 minutes of tDCS stimulation. 3)One day post tDCS treatment. 4)One day post 10 session of back school. 5)Follow up at one month from the back school end.
  Visual analogue scale measure for pain. Score range from 0-10. For rating overall pain: mild = 1-3, moderate = 4-7, severe = 8-10 For rating Chronic Pain: Excellent internal consistency for a single pair of rating between Numeric Pain Rating Scale and Visual Analogue Scale (r = 0.86)

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | 1)One day post tDCS treatment. 2) One day post 10 session of back school. 3) Follow up at one month from the back school end.
  CGI is a scale consisting of two items: the severity of the disease (1=normal, 7=very serious) and the overall improvement (1=much improved, 7=much worse).
Patient Global Assessment (PGA) | 1) One day post tDCS treatment. 2) One day post 10 session of back school. 3) Follow up at one month from the back school end.
  PGA is a scale where the patient gives a score ranging from 1 (serious deterioration) and 7 (big improvement) relative to their pain compared to baseline
Roland Morris Disability Questionnaire (RMDQ) | 1)One day pre-tDCS treatment. 2) One day post tDCS treatment. 3) One day post 10 session of back school. 4) Follow up at one month from the back school end.
  The Roland-Morris disability questionnaire is composed of 24 yes/no questions designed to assess bac 242) Excellent: RMDQ and the Quebec Back Pain Disability Scale (r= 0.77) SIP and RMDQ Assessment The Oswestry Disability Index, the Roland-Morris Disability Questionnaire, and the Quebec Back Pain
The Oswestry Low Back Pain Disability Questionnaire (OLBPDQ) | 1)One day pre-tDCS treatment. 2) One day post tDCS treatment. 3) One day post 10 session of back school. 4) Follow up at one month from the back school end.
Euroquol (Eq-5D) | 1)One day pre-tDCS treatment. 2) One day post tDCS treatment. 3) One day post 10 session of back school. 4) Follow up at one month from the back school end.
The Patient Health Questionnaire - 9 (PHQ-9) | 1)One day pre-tDCS treatment. 2) One day post tDCS treatment. 3) One day post 10 session of back school. 4) Follow up at one month from the back school end.
  PHQ-9 assesses depression symptoms that we tracked as possible confounding factor.
VAS for anxiety (0-10) | 1)One day pre-tDCS treatment. 2) One day post tDCS treatment. 3) One day post 10 session of back school. 4) Follow up at one month from the back school end.
  VAS for anxiety assesses anxiety symptoms that we tracked as possible confounding factor.

CONTACTS AND LOCATIONS:
Locations (1):
- Ferrara University Hospital, Ferrara, Italy